CLINICAL TRIAL: NCT03346356
Title: Evaluation for Implementing the Shaping Healthy Choices Program in the Nevada County 4-H Youth Development Program Utilizing Teenagers as Teachers
Brief Title: SHCP in 4-H Using Teenagers as Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 946461
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Nutrition Knowledge; Vegetable Preferences; Youth Engagement; Civic Responsibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teenagers as cross-age teachers (Experimental): After the initial training, the teenage teachers facilitated the curricula associated with the SHCP, Discovering Healthy Choices and Cooking Up Healthy Choices, approximately twice a month. The curricula can be viewed at http://cns.ucdavis.edu/programs/shcp/curriculum.html. Each activity provided step-by-step instructions that the teenage teachers were asked to follow. Younger youth served as participants for the classroom and garden-based activities.
  Interventions: Behavioral: Teenagers as cross-age SHCP teachers for younger youth
- Comparison group (No Intervention): Youth of similar ages to the intervention group completed the same assessments, but did not receive the intervention.

INTERVENTIONS:
Behavioral: Teenagers as cross-age SHCP teachers for younger youth — Implementation of the SHCP using teenagers as cross-age teachers for younger youth
  Arms: Teenagers as cross-age teachers

SUMMARY:
In close collaboration with the Nevada County 4-H Youth Development Program, the Shaping Healthy Choices Program was implemented utilizing 4-H teenagers as cross-age teachers for younger youth. The 4-H Youth Development Program is an education program of the University of California Cooperative Extension that emphasizes learning citizenship, leadership, and life skills. The program creates positive opportunities for youth to learn, develop skills, and become engaged in their local communities. This is accomplished with combined efforts of youth, volunteer leaders, and University staff and faculty through a fun, hands-on learning approach to non-formal education. As a requirement to participate in the program, all youth had to enroll in 4-H for the 2016-2017 year. Teenagers were initially trained in inquiry-based and experiential learning techniques before facilitating the program. Teenage teachers collectively lead classroom education, garden activities, and cooking demonstrations. Additionally, teenage teachers, UC Cooperative Extension staff, and UC Davis students organized and implemented a community health fair for elementary-aged children.

Measurements were taken on nutrition knowledge, vegetables preferences, civic responsibility, program fidelity, and self-efficacy for teaching nutrition. A parent interview was also conducted to gauge parental engagement and perception of whether their child had behavior changes while participating in the program. Preliminary findings from the parent interview show that children were more likely to support and engage in healthy eating practices throughout their involvement than they had before the program. Children also have expressed interests in continuing their participation in subsequent years. All other data for this intervention are currently undergoing analyses.

ELIGIBILITY:
Inclusion Criteria:

* The research team will recruit and consent youth study participants and their parents from members of the Nevada County 4-H Youth Development Program. Youth study participants must be ages 14-18 for teenage teachers and 8-13 for younger youth participants. Study participants must be able to attend two-hour bimonthly meetings at the 4-H office and/or (depending on the activity) Food Bank garden in Grass Valley, California. Teenage teachers will also be required to complete ten hours of initial training before the start of SHCP implementation. All participants will be required to join the Nevada County 4-H Youth Development Program if they are not already a member. Teenage teachers' registration fees will be paid for by the research team. Comparison youth will be recruited from registered members of the Placer County 4-H Youth Development Program. Placer County 4-H club members will also be ages 14-18 for teenage comparisons and 8-13 for younger youth comparisons.

Exclusion Criteria:

* Foster children and wards of the state will not be enrolled in this study. Children younger than 8 or older than 18 are not eligible to participate.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Change in nutrition knowledge | Change in baseline nutrition knowledge at post-intervention approximately 6 months later
  Nutrition knowledge was assessed using two validated measurement tools: one for younger youth and one for adolescents. Both questionnaires have a similar format and include multiple choice options.

SECONDARY OUTCOMES:
Change in self-efficacy for teaching nutrition | Change in baseline self-efficacy for teaching nutrition at post-intervention approximately 6 months later
  Self-efficacy for teaching nutrition questionnaire includes a questions about competencies for teaching nutrition that are rated using a 5-point Likert scale. This measurement was only used with the teenage teachers.
Change in Civic Responsibility | Change in baseline Civic Responsibility at post-intervention approximately 6 months later
  Civic Responsibility questionnaire measures youth's connection and action within their community using a 6-point Likert scale. This measurement was only used with the teenage teachers.
Change in vegetables preferences | Change in baseline vegetable preferences for teaching nutrition at post-intervention approximately 6 months later
  Vegetables Preferences task involves displaying a whole vegetable as well as a sample of the vegetable for six different vegetables. One-on-one with a research assistant, youth are asked whether they can name the vegetable and a series of application and qualitative questions about that vegetable. This measurement was only used with the younger youth participants.

IPD SHARING:
Plan to Share IPD: No